CLINICAL TRIAL: NCT03232073
Title: Multicenter, Non-comparative Extension of Study AC-058B301, to Investigate the Long-term Safety, Tolerability, and Control of Disease of Ponesimod 20 mg in Subjects With Relapsing Multiple Sclerosis
Brief Title: Long-term Extension to Study AC-058B301 to Investigate Safety, Tolerability and Disease Control of Ponesimod 20 mg in Patients With Relapsing Multiple Sclerosis
Acronym: OPTIMUM-LT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-058B303; AC-058B303 (Other: Janssen Research & Development, LLC); 2016-004719-10 (EudraCT Number)
Record Dates: First submitted 2017-07-20; First posted 2017-07-27 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ponesimod

STUDY DESIGN:
Intervention Model Description: This is a single-group open-label extension study to investigate long-term safety, tolerability and control of disease of ponesimod 20 mg in subjects with RMS. Statistical analyses will be descriptive and therefore all endpoints are exploratory in nature. All exploratory endpoints are listed under primary outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ponesimod (Experimental): 20 mg administered orally once daily
  Interventions: Drug: Ponesimod

INTERVENTIONS:
Drug: Ponesimod — Ponesimod; Film-coated tablet; Oral use. From Day 1 to Day 14, ponesimod is gradually up-titrated until a maintenance dose of 20 mg is reached from Day 15

SUMMARY:
The study AC-058B301 (OPTIMUM; NCT02425644) has been designed to investigate the efficacy, safety and tolerability of ponesimod in subjects with relapsing multiple sclerosis (RMS). The AC-058B303 study is the long-term extension for the core study AC-058B301. The purpose of this long term extension of the core study AC-058B301 is to characterize the long-term safety, tolerability, and control of disease of ponesimod 20 mg in subjects with RMS.

DETAILED DESCRIPTION:
The AC-058B303 study (extension study) is the long-term extension for the AC-058B301 study (core study). The core study has been designed to investigate the efficacy, safety and tolerability of ponesimod in subjects with RMS. The subjects are treated with either ponesimod or the active comparator, teriflunomide in the core study. The purpose of this long term extension of the core study is to characterize the long-term safety and control of disease of ponesimod in subjects with RMS. In particular, the study will allow to observe potential adverse events which may only occur after long term treatment with ponesimod. The study will also investigate the effect of re-initiation of ponesimod after a brief interruption in a relatively large population (all subjects treated with ponesimod in the core study and eligible for the extension study) on disease activity in terms of relapses and MS-related MRI lesions. There is currently limited guidance on when a new MS treatment should be started after discontinuation of teriflunomide and the study will contribute with data on safety and efficacy of switching from teriflunomide to ponesimod after an interruption as mandated by the protocol. The study will also allow confirmation of sustained efficacy of ponesimod in terms of relapses, MRI lesions and reduction of disability accumulation during long-term treatment. In addition, combined data from the core study together with the results of the current extension study will allow comparison of MS activity in subjects who were switched from teriflunomide to ponesimod versus those who were treated with ponesimod in both studies.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Subjects with MS having completed the double-blind treatment in the core study as scheduled
3. Compliance with teriflunomide elimination procedure
4. Women of childbearing potential (WOCBP) must have a negative pre-treatment urine pregnancy test, must agree to undertake 4-weekly urine pregnancy tests, and must have been using reliable methods of contraception. Fertile male subjects participating in the study must agree to use a condom.

Exclusion Criteria:

1. Any of the following cardiovascular conditions on Day 1 pre-dose:

   1. Resting heart rate (HR) < 50 bpm;
   2. Presence of second degree atrioventricular (AV) block or third degree AV block or a QTcF interval > 470 ms (females), > 450 ms (males);
2. Any of the following alerts from central laboratory at Visit 14 of the core study (EOT) which was confirmed as an alert at repeated testing or not repeated prior to FU1 of the core study:

   1. Lymphocyte count: < 0.2 x 109/L;
   2. Neutrophil count <1.0 × 109/L;
   3. Platelet count < 50 × 109/L;
   4. Creatinine clearance < 30 mL/min
3. At Visit 14 of the core study (EOT) >30% decrease from core study baseline FEV1 and/or FVC;
4. Clinically significant, persistent respiratory AEs (e.g., dyspnea) not resolved prior to first dosing in the extension study.
5. Macular edema at any time between Visit 1 (Screening) in the core study and Day 1 of the extension study.
6. Presence of the following at core study Visit 14 (EOT, Week 108), FU1, or abbreviated visit FU2, or on Day 1 of the extension study pre-dose:

   1. Suspected opportunistic infection of the CNS or any other infection which, in the opinion of the investigator, contraindicates re-start of the study drug;
   2. Stevens-Johnson syndrome or toxic epidermal necrolysis or drug reaction with eosinophilia and systemic symptoms.
7. Need for and intention to administer forbidden study treatment-concomitant therapy
8. Women who are pregnant or lactating.
9. Male subjects wishing to parent a child;
10. Treatment with any MS Disease Modifying Therapies;
11. Any other clinically relevant medical or surgical condition, which, in the opinion of the investigator, would put the subject at risk by participating in the study;
12. Subjects unlikely to comply with the extension study protocol based on investigator best judgment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 877 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Sidorenko, MD, PhD, Study Director — Actelion
Locations (148):
- United States (9):
  - The Research Center of Southern California, LLC, Carlsbad, California
  - The Neurology Group, Pomona, California
  - Mountain View Clinical Research, Denver, Colorado
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - University of South Florida, Tampa, Florida
  - Josephson Wallack Munshower Neurology, PC, Indianapolis, Indiana
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Ohio Health, Columbus, Ohio
  - Advanced Neurosciences Institute, Franklin, Tennessee
- Belarus (5):
  - Grodno University Hospital, Grodno
  - Minsk City Clinical Hospital 5, Minsk
  - Republican Scientific Clinical Centre, Minsk
  - Vitebsk Regional Diagnostic Center, Vitebsk
  - Vitebsk Regional Clinical Hospital, Vitebsk
- University Clinicl Center Sarajevo, Sarajevo, Bosnia and Herzegovina
- Bulgaria (7):
  - UMHAT Sveti Georgi, Plovdiv
  - Multiprofile Hospital for Active Treatment in Neurology and Psychiatry Sveti Naum, Sofia
  - Multiprofile Hospital For Active Treatment National Cardiology Hospital, Ead, Sofia
  - Acibadem City Clinic Tokuda Hospital, Sofia
  - St Ivan Rilski University Multiprofile Hospital For Active Treatment, Sofia
  - University Multiprofile Hospital for Active Treatment Alexandrovska EAD, Sofia
  - Military Medical Academy Multiprofile Hospital for Active Treatment Sofia, Sofia
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Ottawa Hospital, Ottawa, Ontario
  - Recherche Sepmus Inc., Greenfield Park, Quebec
- Croatia (2):
  - Ch Osijek, Osijek
  - University Hospital Center Zagreb, Zagreb
- Czechia (8):
  - Fakultní nemocnici Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Nemocnice Jihlava, Jihlava
  - Fakultni Nemocnice Ostrava, Ostrava-Poruba
  - Pardubicka krajska nemocnice a s, Pardubice
  - Vseobecna Fakultní Nemocnice, Prague
  - FN Motol, Prague
  - Krajska zdravotni, a.s. - Nemocnice Teplice, o.z., Teplice
- Finland (2):
  - Suomen Terveystalo Tampere, Tampere
  - Mehilainen NEO, Turku
- France (5):
  - Hopital Pellegrin CHU Bordeaux, Bordeaux
  - CHU Clermont-Ferrand - Hopital Gabriel Montpied, Clermont-Ferrand
  - Hopital Nord Laennec CHU NANTES, Nantes
  - Hopital PASTEUR, Nice
  - Nouvel Hopital Civil, Strasbourg
- Georgia (5):
  - LTD 'Aversi Clinic', Tbilisi
  - P. Sarajishvili Institute of Neurology, Tbilisi
  - Pineo Medical Ecosystem Ltd, Tbilisi
  - S.Khechinashvili University Hospital, Tbilisi
  - Curatio, Jsc, Tbilisi
- Germany (4):
  - Universitätsklinikum Carl-Gustav-Carus Dresden, Dresden
  - Helios Klinikum Erfurt, Erfurt
  - Panakeia - Arzneimittelforschung GmbH, Leipzig
  - Universitatsmedizin der Johannes Gutenberg Universitat Mainz, Mainz
- Greece (3):
  - 401 Military Hospital, Athens
  - Naval Hospital of Athens, Athens
  - Medical Center of Athens, Marousi
- Hungary (5):
  - Uzsoki Utcai Korhaz, Budapest
  - Jahn Ferenc Del-pesti Korhaz es Rendelointezet, Budapest
  - Valeomed EGÉSZSÉGÜGYI KÖZPONT, Esztergom
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Kistarcsai Flor Ferenc Korhaz, Kistarcsa
- Israel (4):
  - Barzilai Medical Center, Ashkelon
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Ziv Medical Center, Safed
- Italy (2):
  - Ospedale San Salvatore, L’Aquila
  - Azienda Ospedaliera Sant Andrea, Roma
- Latvia (3):
  - Pauls Stradins Clinical University Hospital, Riga
  - Latvias Juras medicinas centrs Ltd, Riga
  - Rīgas Austrumu klīniskā universitātes slimnīca, Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - VsI Respublikine Siauliu ligonine, V., Šiauliai
- Mexico (2):
  - Unidad de Investigacion En Salud, Chihuahua City
  - CRI Centro Regiomontano de Investigacion SC, Nuevo León
- Poland (11):
  - Neurocentrum Bydgoszcz Sp Z O O, Bydgoszcz
  - Copernicus Podmiot Leczniczy Sp. z o.o, Gdansk
  - Neuro Centrum Centrum Terapii SM, Katowice
  - NEURO MEDIC Janusz Zbrojkiewicz Poradnia Wielospecjalistyczna, Katowice
  - Centrum Kompleksowej Rehabilitacji, Konstancin-Jeziorna
  - Centrum Opieki Zdrowotnej Orkan Med, Ksawerów
  - Indywidualna Praktyka Lekarska Prof. Konrad Rejdak, Lublin
  - Szpital Kliniczny im Heliodora Swiecickiego Uniwersytetu Medycznego im Karola Marcinkowskiego w Po, Poznan
  - Clinical Research Center sp z o o MEDIC R s k, Poznan
  - NZOZ NEURO KARD Ilkowski i Partnerzy Sp Partnerska Lekarzy, Poznan
  - WroMedica I Bielicka A Strzalkowska s c, Wroclaw
- Portugal (4):
  - Hospital de Braga, Braga
  - Hospitais da universidade de Coimbra, Coimbra
  - Hosp. Cuf Descobertas, Lisbon
  - H. Santo António - Centro Hospitalar do Porto, Porto
- Romania (4):
  - Spitalul Universitar de Urgenta Militar Central 'Dr. Carol Davila', Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Spitalul Clinic Judetean de Urgenta Pius Brinzeu, Timișoara
- Russia (26):
  - Barnaul Territorial Clinical Hospital, Barnaul
  - St. Joseph Belgorod Regional Hospital, Belgorod
  - Bryansk Regional Hospital #1, Bryansk
  - Research Medical Center Your Health, Kazan'
  - Federal State Budgetary Institution, Krasnoyarsk
  - State Budgetary Healthcare Institution Kursk Region Kursk Regional Clinical Hospital, Kursk
  - Clinical City Hospital #1, Moscow
  - State Health Care Institution Of Moscow, Moscow
  - Central Clinical Hospital N.A.Semashko, Moscow
  - Municipal Clinical Hospital # 3, Nizhny Novgorod
  - Siberian District Medical Center of Federal Medical-Biological Agency, Novosibirsk
  - Federal Scientific Clinical Center of Physico-Chemical Medicine, Odintsovo
  - Perm State Medical Academy n.a. E. A. Vagner, Perm
  - City Clinical Hospital # 2, Pyatigorsk
  - Municipal Multi-Specialty Hospital # 2, Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - City Clinical Hospital #31, Saint Petersburg
  - Institute of Human Brain Ras, Saint Petersburg
  - City Hospital# 40, Saint Petersburg
  - State Healthcare Institution Samara Regional Clinical Hospital named after V.D.Seredavin, Samara
  - Smolensk Regional Clinical Hospital, Smolensk
  - Siberian State Medical University, Tomsk
  - Tver Regional Clinical Hospital, Tver'
  - GUZ Novgorod Regional Clinical Hospital, Veliky Novgorod
  - Yaroslavl Clinical Hospital #8, Yaroslavl
  - Sverdlovsk Region Clinical Hospital #1, Yekaterinburg
- Serbia (4):
  - Clinical Hospital Center Zvezdara, Belgrade
  - Vojnomedicinska Akademija, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - University Clinical Center NIS, Niš
- Spain (7):
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Vithas Nisa Sevilla, Seville
- Sweden (2):
  - Sahlgrenska Universitetsjukhuset, Gothenburg
  - Centrum för Neurologi, Stockholm
- Karadeniz Teknik University Medical Faculty, Trabzon, Turkey (Türkiye)
- Ukraine (14):
  - Public Non-profit Enterprise: Chernihiv City Hospital #4 under Chernihiv City Council, Chernihiv
  - Municipal health care institution Chernihiv Regional Hospital, Chernihiv
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - Limited Liability Company 'Neuro Global', Ivano-Frankivsk
  - Kharkiv Railway Clinical Hospital N1 Of Brance 'Health Center', Kharkiv
  - Kharkiv Postgrad Academy, Dept of Neurology #1 At Hosp #7, Kharkiv
  - National Research Center for Radiation Medicine, Kyiv
  - Public Non-Profit Enterprise: Lviv City Clinical Hospital #5, Lviv
  - Lviv Clinical Regional Hospital, Lviv
  - Odessa National Medical University, Odesa
  - ME 'Poltava Regional Clinical Hospital n.a. M.V. Sklifosovsky of the Poltava Regional Council', Poltava
  - Mnce 'Ternopil Regional Clinical Psychoneurology Hospital' of Trb, Ternopil
  - Medical Center Salutem LLC, Vinnytsia
  - O.F. Herbachevskyi Regional Clinical Hospital, Zhytomyr
- United Kingdom (2):
  - Royal Preston Hospital, Preston
  - Salford Royal NHS Foundation Trust, Salford

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 877 participants entered this extension study from the core study (NCT02425644) and all received at least one dose of ponesimod 20 milligrams (mg) treatment.
Pre-assignment Details: Efficacy data: presented for extension set (ES; who consented and had 1 dose of ponesimod in extension study) in combined analysis period (included all available data from randomization in core study up to extension end of study [EOS] for those who entered ES). Safety data: presented for ES in extension analysis period (included all available data collected on or after date of 1st intake of ponesimod in extension study, through last treatment date in extension study+15 days).
Groups:
- Ponesimod 20 mg (Core and Extension Study): Participants with multiple sclerosis (MS) who were treated with ponesimod 20 milligrams (mg) in the core study (NCT02425644), and entered into this extension study, received a 14-day gradual up-titrated treatment (from 2 mg to 10 mg) of ponesimod tablet orally once daily from Days 1 to 14. Participants received a daily maintenance dose of ponesimod 20 mg tablet orally once daily from Day 15 up to Week 240 or till ponesimod became commercially available in a participant's country. Participants located in Ukraine had an extended treatment duration up to 288 weeks in the extension study due to the regional crisis.
- Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension): Participants with multiple sclerosis (MS) who were treated with teriflunomide 14 mg in the core study (NCT02425644), and entered into this extension study, received a 14-day gradual up-titrated treatment (from 2 mg to 10 mg) of ponesimod tablet orally once daily from Days 1 to 14. Participants received a daily maintenance dose of ponesimod 20 mg tablet orally once daily from Day 15 up to Week 240 or till ponesimod became commercially available in a participant's country. Participants located in Ukraine had an extended treatment duration up to 288 weeks in the extension study due to the regional crisis.
Period: Overall Study
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Started | 439 | 438
Completed | 352 | 371
Not Completed | 87 | 67
Not completed — Death | 1 | 0
Not completed — Adverse Event | 7 | 12
Not completed — Lost to Follow-up | 6 | 6
Not completed — Lack of Efficacy | 10 | 8
Not completed — Physician Decision | 9 | 2
Not completed — Withdrawal by Subject | 54 | 39

BASELINE CHARACTERISTICS:
Population: The extension set included all participants who signed an informed consent to enter the extension study and who received at least one dose of ponesimod study medication in the extension study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension) | Total
Number analyzed (Participants) | 439 | 438 | 877
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 439 | 438 | 877
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (8.75) | 37.2 (8.75) | 36.8 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 286 | 290 | 576
  Male | 153 | 148 | 301
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 17 | 39
  Not Hispanic or Latino | 409 | 411 | 820
  Unknown or Not Reported | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 429 | 430 | 859
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Annualized Confirmed Relapse Rate (ARR)
Description: ARR: number of confirmed relapses per patient-year. Relapse: new, worsening, or recurrent neurological symptoms that occurred at least 30 days after the onset of a preceding relapse, and that lasted at least 24 hours, in the absence of fever or infection. A confirmed relapse is identified when a patient's symptoms worsen as indicated by an increase in their Expanded Disability Status Scale (EDSS) or Functional Systems (FS) scores, consistent with previous clinically stable assessments. Specific criteria for a confirmed relapse include: An increase of 0.5 points on EDSS; (unless EDSS=0, then requires an increase of 1.0-point); An increase of at least 1.0 point in at least two FS scores; or a 2.0-point increase in one FS score (excluding bladder/bowel and cerebral). Rating individual FS scores is used to rate EDSS along with observations and information concerning gait and use of assistance. EDSS is ordinal clinical rating scale ranging:0 (normal)-10 (death due to MS).
Time Frame: From randomization in the core study up to the end of study (EOS) in the extension study. The actual time varied for each participant and could be up to 98.5 months
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: relapses per patient-year
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 439 | 438
relapses per patient-year | 0.143 [0.123 to 0.167] | 0.184 [0.158 to 0.213]
Statistical Analysis 1: Comparison: Ponesimod 20 mg (Core and Extension Study) vs Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension); Test type: Superiority; Treatment Effect (Rate Ratio) = 0.779, 95% CI [0.629 to 0.965]

2. Primary Outcome: Time From Core Study Randomization to First Confirmed Relapse
Description: Time to first confirmed relapse: date of first confirmed relapse (in either core or extension study) minus date of randomization in core study+1 day. Relapse: new, worsening, or recurrent neurological symptoms that occurred at least 30 days after the onset of a preceding relapse, and that lasted at least 24 hours in absence of fever or infection. A confirmed relapse: when patient's symptoms worsen as indicated by an increase in their EDSS/FS scores, consistent with previous clinically stable assessments. Specific criteria for confirmed relapse are: An increase of 0.5 points on EDSS; (unless EDSS=0, then requires an increase of 1.0-point); An increase of at least 1.0 point in at least two FS scores; or a 2.0-point increase in one FS score (excluding bladder/bowel and cerebral). Rating individual FS scores is used to rate EDSS along with observations and information concerning gait and use of assistance. EDSS is ordinal clinical rating scale ranging:0(normal)-10(death due to MS).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 439 | 438
Weeks | 402.71 [82.29 to NA] — NA refers to data for inter-quartile upper limit which was not estimable to due to low number of events. | NA [53.57 to NA] — NA refers to data for median and inter-quartile upper limit which were not estimable to due to low number of events.

3. Primary Outcome: Time to First 12-week Confirmed Disability Accumulation (CDA)
Description: Time to first 12-week CDA is defined as start date of the first 12-week CDA minus date of randomization in the core study + 1 day. A 12-week CDA is defined as a 12-week sustained increase from the core baseline EDSS score, which is confirmed at a scheduled visit after 12-weeks. CDA is defined as: (a) Sustained increase of at least 1.5 in EDSS for participants with a core baseline EDSS score of 0; (b) Sustained increase of at least 1.0 in EDSS for participants with a core baseline EDSS score of 1.0 to 5.0; (c) Sustained increase of at least 0.5 in EDSS for participants with a core baseline EDSS score >=5.5, confirmed after 12 weeks. EDSS is an ordinal clinical rating scale ranging from 0 (normal neurological examination) to 10 (death due to MS). Core baseline for efficacy: last non-missing value recorded before or on randomization in the core study for each outcome measure and participant individually.
Time Frame: From baseline in the core study up to the end of study (EOS) in the extension study. The actual time varied for each participant and could be up to 98.5 months
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 439 | 438
Weeks | NA [NA to NA] — NA refers to data for median, inter-quartile lower and upper limit which were not estimable to due to low number of events. | NA [254.86 to NA] — NA refers to data for median and inter-quartile upper limit which were not estimable to due to low number of events.

4. Primary Outcome: Time to First 24-week Confirmed Disability Accumulation (CDA)
Description: Time to first 24-week CDA was defined as start date of the first 24-week CDA minus date of randomization in the core study + 1 day. A 24-week CDA was defined as a 24-week sustained increase from the core baseline EDSS score, which is confirmed at a scheduled visit after 24-weeks. CDA was defined as: (a) Sustained increase of at least 1.5 in EDSS for participants with a core baseline EDSS score of 0; (b) Sustained increase of at least 1.0 in EDSS for participants with a core baseline EDSS score of 1.0 to 5.0; (c) Sustained increase of at least 0.5 in EDSS for participants with a core baseline EDSS score >=5.5, confirmed after 24 weeks. EDSS was an ordinal clinical rating scale ranging from 0 (normal neurological examination) to 10 (death due to MS). Core baseline for efficacy: last non-missing value recorded before or on randomization in the core study for each outcome measure and participant individually.
Time Frame: as for outcome 3
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 439 | 438
Weeks | NA [NA to NA] — NA refers to data for median, inter-quartile lower and upper limit which were not estimable to due to low number of events. | NA [313.29 to NA] — NA refers to data for median and inter-quartile upper limit which were not estimable to due to low number of events.

5. Primary Outcome: Percentage of Participants With Absence of Relapses
Description: Relapse: new, worsening, or recurrent neurological symptoms that occurred at least 30 days after the onset of a preceding relapse, and that lasted at least 24 hours in absence of fever or infection. A confirmed relapse: when patient's symptoms worsen as indicated by an increase in their EDSS/FS scores, consistent with previous clinically stable assessments. Specific criteria for confirmed relapse: An increase of 0.5 points on EDSS; (unless EDSS=0, then requires an increase of 1.0-point); An increase of at least 1.0 point in at least two FS scores; or a 2.0-point increase in one FS score (excluding bladder/bowel and cerebral). Rating individual FS scores is used to rate EDSS along with observations and information concerning gait and use of assistance. EDSS is ordinal clinical rating scale ranging:0(normal)-10(death due to MS). Core baseline for efficacy: last non-missing value recorded before or on randomization in the core study for each outcome measure and participant individually.
Time Frame: as for outcome 3
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 439 | 438
Percentage of Participants | 56.7 | 51.6

6. Primary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS)
Description: EDSS is ordinal clinical rating scale based on standard neurological examination for assessing neurological disability and impairment in MS. Seven FS scores were rated on a scale ranged from 0 to 5 or 6 to assess visual, brain, stem, pyramidal, cerebellar, sensory, bowel and bladder, and cerebral functions while ambulation was scored on scale ranged from 0 to 12 to assess walking distance and assistance. Individual FS scores were then used in conjugation with ambulation score to obtain EDSS score which ranged from 0 (normal) to 10 (death due to MS) in 0.5 unit increments that represented higher levels of disability. Core baseline for efficacy is defined as the last non-missing value recorded before or on randomization in the core study for each outcome measure and each participant individually.
Time Frame: as for outcome 3
Population: The extension set included all participants who signed an informed consent to enter the extension study and who received at least one dose of ponesimod study medication in the extension study. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 346 | 364
Score on a scale | 0.16 (1.008) | 0.34 (1.105)

7. Primary Outcome: Percentage of Participants With No Evidence of Disease Activity (NEDA) Status According to NEDA With Three Components (NEDA-3) at Extension End of Study
Description: NEDA-3 up to extension EOS is defined by the absence of confirmed relapse, gadolinium-enhancing (Gd+ T1) lesions, new or enlarging T2 lesions, and 12-week CDA. If at least one of the criteria was not fulfilled or the participant discontinued treatment prematurely, the participant was not considered to have achieved NEDA-3. Confirmed relapse: when patient's symptoms worsen as indicated by an increase in their EDSS/FS scores, consistent with previous clinically stable assessments. Rating individual FS scores is used to rate EDSS along with observations and information concerning gait and use of assistance. EDSS is ordinal clinical rating scale ranging: 0 (normal)-10 (death due to MS). Core baseline for efficacy is defined as the last non-missing value recorded before or on randomization in the core study for each outcome measure and each participant individually.
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 439 | 436
Percentage of Participants | 17.5 | 7.5

8. Primary Outcome: Percentage of Participants With No Evidence of Disease Activity (NEDA) Status According to NEDA With Four Components (NEDA-4) at Extension End of Study
Description: NEDA-4 up to EOS is defined by the absence of confirmed relapse, Gd+ T1 lesions, new or enlarging T2 lesions, 12-week CDA until EOS, and absence of annual brain volume decrease >=0.4% from core baseline up to extension EOS. If at least one of the criteria was not fulfilled or the participant discontinued treatment prematurely, the participant was not considered to have achieved NEDA-4. Confirmed relapse: when patient's symptoms worsen by an increase in their EDSS/FS scores, consistent with previous clinically stable assessments. Rating individual FS scores is used to rate EDSS along with observations and information concerning gait and use of assistance. EDSS is ordinal clinical rating scale ranging: 0 (normal)-10 (death due to MS). Core baseline for efficacy is defined as the last non-missing value recorded before or on randomization in core study for each outcome measure and each participant individually.
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 437 | 435
Percentage of Participants | 5.2 | 2.3

9. Primary Outcome: Percent Change From Baseline in Brain Volume (PCBV) Measured by Magnetic Resonance Imaging (MRI)
Description: Percent change from baseline in brain volume (PCBV) measured by MRI were reported. Normalized Brain Volume at core baseline was measured in cubic centimeter (cm^3). Core baseline for efficacy is defined as the last non-missing value recorded before or on randomization in the core study for each outcome measure and each participant individually. In this outcome measure, results were presented for extension end of treatment visit.
Time Frame: From baseline in the core study up to the end of treatment (EOT) in the extension study. The actual time varied for each participant and could be up to 94.8 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 196 | 193
Percent Change | -2.52 (2.179) | -2.72 (2.024)

10. Primary Outcome: Cumulative Number of Combined Unique Active Lesions (CUAL) Measured by MRI
Description: CUALs was calculated as sum of new T1 Gadolinium-enhanced (Gd+) lesions and new or enlarging T2 lesions (without double-counting of lesions) from baseline up to extension EOS based on the Magnetic resonance imaging (MRI). Average number of lesions per patient-year were reported. Results are based on a negative-binomial regression model. Core baseline for efficacy is defined as the last non-missing value recorded before or on randomization in the core study for each outcome measure and each participant individually.
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: CUAL per patient-year
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 438 | 435
CUAL per patient-year | 1.352 [1.153 to 1.586] | 1.954 [1.667 to 2.291]

11. Primary Outcome: Number of Gadolinium-enhancing (Gd+) T1 Lesions Measured by MRI
Description: Number of Gd+ T1 lesions measured by MRI were reported. Results are based on a negative-binomial regression model. Core baseline for efficacy is defined as the last non-missing value recorded before or on randomization in the core study for each outcome measure and each participant individually. For this outcome measure, results presented here are for the Extension end-of-treatment visit.
Time Frame: as for outcome 9
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: Gd+ T1 lesions
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 350 | 347
Gd+ T1 lesions | 0.211 [0.131 to 0.341] | 0.395 [0.250 to 0.622]

12. Primary Outcome: Cumulative Number of New or Enlarging T2 Lesions Measured by MRI
Description: Cumulative number of new or enlarging T2 lesions measured by MRI were reported. Average number of lesions per year were reported. Results are based on a negative-binomial regression model. Core baseline for efficacy is defined as the last non-missing value recorded before or on randomization in the core study for each outcome measure and each participant individually.
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: Lesions per year
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 438 | 435
Lesions per year | 1.352 [1.152 to 1.586] | 1.951 [1.664 to 2.287]

13. Primary Outcome: Change From Baseline in Volume of MRI Lesions (T2 Lesions and T1 Hypointense Lesions)
Description: Change from baseline in volume of MRI lesions (T2 lesions, T1 hypointense lesions) were reported. Core baseline for efficacy is defined as the last non-missing value recorded before or on randomization in the core study for each outcome measure and each participant individually. In this outcome measure, results were presented for extension end of treatment visit.
Time Frame: as for outcome 9
Population: The extension set included all participants who signed an informed consent to enter the extension study and who received at least one dose of ponesimod study medication in the extension study. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here, 'n' (number analyzed) is defined as participants analyzed at specified categories.
Measure: Mean (Standard Deviation); unit: cubic millimeters (mm^3)
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 347 | 348
cubic millimeters (mm^3)
  T2 Lesions | -435.7 (2822.71) | 91.5 (3647.08)
  T1 Hypointense Lesions: number analyzed (Participants) | 346 | 345
  T1 Hypointense Lesions | 165.6 (1427.30) | 309.4 (1712.36)

14. Primary Outcome: Number of Participants With Absence of MRI Lesions (Gd+ T1 Lesions, New or Enlarging T2 Lesions)
Description: Number of participants with absence of MRI lesions (Gd+ T1 lesions, new or enlarging T2 lesions) were reported. Core baseline for efficacy is defined as the last non-missing value recorded before or on randomization in the core study for each outcome measure and each participant individually. In this outcome measure, results were presented for extension end of treatment visit.
Time Frame: as for outcome 9
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 439 | 435
Participants
  Gd+ T1 lesions | 293 | 236
  T2 lesions: number analyzed (Participants) | 438 | 435
  T2 lesions | 152 | 101

15. Primary Outcome: Percentage of Gd+ Lesions at Baseline Evolving to Persistent Black Holes (PBHs)
Description: Percentage of Gd+ lesions at baseline evolving to PBHs were reported. Core baseline for efficacy is defined as the last non-missing value recorded before or on randomization in the core study for each outcome measure and each participant individually. In this outcome measure, results were presented for extension end of treatment visit.
Time Frame: as for outcome 9
Population: as for outcome 6
Measure: Number; unit: Percentage of lesions
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 350 | 346
Percentage of lesions | 22.3 | 25.1

16. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs were reported. An AE is any untoward medical event that occurs in a participants being administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs are defined as AEs occurring from start of treatment up to treatment end date + 15 days.
Time Frame: From the start of study treatment in the extension study up to the end of study treatment + 15 days in the extension study. The actual time varied for each participant and could be up to 71.8 months + 15 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 439 | 438
Participants | 411 | 410

17. Primary Outcome: Number of Participants With Treatment-emergent New Morphological Electrocardiogram (ECG) Abnormalities
Description: Number of participants with treatment-emergent new morphological ECG abnormalities were reported. Treatment-emergent new morphological ECG abnormalities are defined as those ECG abnormalities occurring from start of treatment up to treatment end date + 15 days.
Time Frame: as for outcome 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 439 | 438
Participants | 153 | 140

18. Primary Outcome: Actual Values of 12-lead ECG Measurements up to End of Study Treatment: Heart Rate
Description: Actual values of 12-lead ECG measurements up to end of study treatment: heart rate were reported. In this outcome measure, results were presented for extension end of treatment visit.
Time Frame: From the start of study treatment in the extension study up to the end of study treatment in the extension study. The actual time varied for each participant and could be up to 71.8 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 361 | 361
Beats per minute (bpm) | 67.4 (9.64) | 67.6 (9.33)

19. Primary Outcome: Actual Values of 12-lead ECG Measurements up to End of Study Treatment: PR, QRS, QT, QTcB, QTcF
Description: Actual values of 12-lead ECG measurements up to end of study treatment: PR, QRS, QT, QTcB, QTcF were reported. In this outcome measure, results were presented for extension end of treatment visit.
Time Frame: as for outcome 18
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: millisecond (ms)
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 361 | 361
millisecond (ms)
  PR Interval | 150.0 (20.41) | 153.3 (20.27)
  QRS Duration | 92.1 (9.22) | 93.3 (10.63)
  QT Interval | 392.5 (27.26) | 391.0 (25.67)
  QTcB Interval | 414.8 (19.20) | 413.8 (19.66)
  QTcF Interval | 406.9 (17.78) | 405.7 (17.78)

20. Primary Outcome: Change in Heart Rate (HR) From Baseline up to End of Study Treatment
Description: Change in heart rate (HR) from baseline up to end of study treatment were reported.
Time Frame: as for outcome 18
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 361 | 361
beats per minute (bpm) | -1.7 (10.00) | -1.5 (9.17)

21. Primary Outcome: Change in PR, QRS, QT, QTcB, QTcF From Baseline up to End of Study Treatment
Description: Change in PR, QRS, QT, QTcB, QTcF from baseline up to end of study treatment were reported.
Time Frame: as for outcome 18
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: millisecond (ms)
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 361 | 361
millisecond (ms)
  PR Interval | 0.5 (14.09) | 2.0 (14.37)
  QRS Duration | -0.4 (6.79) | 2.9 (6.88)
  QT Interval | 7.8 (25.68) | 8.9 (21.66)
  QTcB Interval | 2.9 (16.75) | 5.2 (17.07)
  QTcF Interval | 4.6 (15.28) | 6.5 (14.18)

22. Primary Outcome: Absolute Values in Forced Expiratory Volume in 1 Second (FEV1) and Forced Vital Capacity (FVC) Values
Description: Absolute values in FEV1 and FVC values were reported. FEV1: the maximal volume of air exhaled from the lungs in 1 second of a forced expiration from a position of full inspiration as measured by spirometer. FVC: the volume of air (in liters) that can be forcibly blown out after full inspiration in the upright position. Extension baseline for safety is the last valid non-missing assessment that is taken on or after EOT visit in the core study, and prior to first study drug intake in the extension study. Results are presented for extension end of treatment visit.
Time Frame: From extension study baseline up to the end of study treatment in the extension study. The actual time varied for each participant and could be up to 71.8 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 315 | 327
Liters (L)
  FEV1 | 3.01 (0.768) | 3.08 (0.797)
  FVC | -3.96 (0.965) | 4.04 (1.031)

23. Primary Outcome: Percent Change in (FEV1) and Forced Vital Capacity (FVC) From Baseline (%)
Description: Percent change in FEV1 and FVC from baseline (%) were reported. FEV1: the maximal volume of air exhaled from the lungs in 1 second of a forced expiration from a position of full inspiration as measured by spirometer. FVC: the volume of air (in liters) that can be forcibly blown out after full inspiration in the upright position. Extension baseline for safety is the last valid non-missing assessment that is taken on or after EOT visit in the core study, and prior to first study drug intake in the extension study. In this outcome measure, results were presented for extension end of treatment visit.
Time Frame: as for outcome 22
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 315 | 327
Percent change
  FEV1 | -7.96 (13.356) | -6.75 (12.323)
  FVC | -5.09 (11.793) | -3.93 (12.141)

24. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAEs)
Description: Number of participants with treatment-emergent SAEs were reported. A SAE was defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, leads to a congenital anomaly/birth defect in the offspring of a participant, or was an important medical event. Treatment-emergent SAEs are defined as SAEs occurring from start of treatment up to treatment end date + 15 days.
Time Frame: as for outcome 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 439 | 438
Participants | 56 [lower limit 0.442] | 57 [lower limit 0.380]

25. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events of Special Interest (AESIs)
Description: Number of participants with treatment-emergent AESIs were reported. AESIs included bradyarrhythmia occurred post-first dose, macular edema, bronchoconstriction, severe liver injury, serious opportunistic infections including progressive multifocal leukoencephalopathy (PML), skin cancer, non-skin malignancy, convulsions, unexpected neurological or psychiatric symptoms/signs (posterior reversible encephalopathy syndrome [PRES], acute disseminated encephalomyelitis [ADEM], and atypical MS relapses). Treatment-emergent AESIs are defined as AESIs occurring from start of treatment up to treatment end date + 15 days.
Time Frame: as for outcome 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 439 | 438
Participants
  Bradyarrhythmia occurring post-first dose | 11 | 13
  Severe liver injury | 5 | 5
  Bronchoconstriction | 31 | 25
  Macular edema | 4 | 6
  Serious opportunistic infections including PML | 2 | 1
  Skin cancer | 4 | 3
  Non-skin malignancy | 4 | 3
  Unexpected neurological or psychiatric symptoms / signs (PRES, ADEM, atypical MS relapses) | 1 | 2
  Convulsions | 2 | 3

26. Primary Outcome: Number of Participants With AE Leading to Premature Discontinuation of Study Treatment
Description: Number of participants with AE leading to premature discontinuation of study treatment were reported. An AE is any untoward medical event that occurs in a participant being administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs are defined as AEs occurring from start of treatment up to treatment end date + 15 days.
Time Frame: as for outcome 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 439 | 438
Participants | 34 | 41

27. Primary Outcome: Number of Participants With Treatment-emergent Decrease From Baseline >20% and >30% in FEV1 or FVC
Description: Number of participants with treatment-emergent decrease from baseline >20% and >30% in FEV1 or FVC were reported. Treatment-emergent is defined as events occurring from start of treatment up to treatment end date + 15 days (that is, findings not present at any assessment prior to first treatment in the extension study).
Time Frame: as for outcome 16
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 424 | 423
Participants
  FEV1: >20 % | 80 | 82
  FEV1: >30 % | 18 | 21
  FVC: >20 % | 54 | 60
  FVC: >30 % | 19 | 15

28. Primary Outcome: Number of Participants With Treatment-emergent Decrease of >20% Points in Percent Predicted FEV1 and FVC From Baseline
Description: Number of participants with treatment-emergent decrease of >20% points in percent predicted FEV1 and FVC from baseline were reported. Treatment-emergent is defined as events occurring from start of treatment up to treatment end date + 15 days (that is, findings not present at any assessment prior to first treatment in the extension study).
Time Frame: as for outcome 16
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 423 | 423
Participants
  FEV1: >20 % | 70 | 68
  FVC: >20 % | 59 | 57

29. Primary Outcome: Number of Participants With a Decrease of >=200 mL or >=12% in FEV1 or FVC From Baseline to EOT
Description: Number of participants with a decrease of >=200 mL or >=12% in FEV1 or FVC from baseline to EOT were planned to be reported. Extension baseline for safety is the last valid non-missing assessment that is taken on or after EOT visit in the core study, and prior to first study drug intake in the extension study. This endpoint is not relevant as a substantial proportion of patients continued onto post-treatment disease-modifying therapy (DMT), hence it cannot provide an assessment of reversibility.
Time Frame: as for outcome 22
Population: as for baseline characteristics
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 0 | 0

30. Primary Outcome: Change in FEV1 and FVC (% Predicted) From Baseline to End of Treatment (EOT)
Description: Change in FEV1 and FVC (% predicted) from baseline to EOT were predicted. Extension baseline for safety is the last valid non-missing assessment that is taken on or after EOT visit in the core study, and prior to first study drug intake in the extension study.
Time Frame: as for outcome 22
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage predicted change
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 315 | 327
Percentage predicted change
  FEV1 | -7.14 (13.315) | -5.43 (11.839)
  FVC | -4.70 (13.129) | -3.19 (13.081)

31. Primary Outcome: Change in FEV1 and FVC (% Predicted) From Baseline to End of Study (EOS)
Description: Change in FEV1 and FVC (% predicted) from baseline to EOS were predicted. Extension baseline for safety is the last valid non-missing assessment that is taken on or after EOT visit in the core study, and prior to first study drug intake in the extension study.
Time Frame: From extension study baseline up to the end of study in the extension study. The actual time varied for each participant and could be up to 73.2 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage predicted change
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 288 | 299
Percentage predicted change
  FEV1 | -5.95 (12.854) | -4.08 (14.365)
  FVC | -4.48 (13.727) | -1.98 (15.747)

32. Primary Outcome: Absolute Change in Lung Diffusion Capacity as Assessed by Diffusing Capacity for the Lungs Measured Using Carbon Monoxide (DL[CO]) From Baseline
Description: Absolute change in lung diffusion capacity as assessed by DL[CO] from baseline were reported. Extension baseline for safety is the last valid non-missing assessment that is taken on or after EOT visit in the core study, and prior to first study drug intake in the extension study.
Time Frame: as for outcome 31
Population: The DL[CO] sub-study extension set included all participants in the extension set who have consented to participate in the DL[CO] sub-study during the extension study. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Millimoles/minute/kilopascal
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 65 | 53
Millimoles/minute/kilopascal | 0.7 (3.44) | 0.1 (4.17)

33. Primary Outcome: Change in DL[CO] (% Predicted) From Baseline to EOT
Description: Change in DL[CO] (% predicted) from baseline to EOT were predicted. Extension baseline for safety is the last valid non-missing assessment that is taken on or after EOT visit in the core study, and prior to first study drug intake in the extension study.
Time Frame: as for outcome 22
Population: The DL[CO] sub-study extension set includes all participants in the extension set who have consented to participate in the DL[CO] sub-study during the extension study. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage predicted DL[CO]
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 50 | 41
Percentage predicted DL[CO] | 5.7 (32.20) | -9.4 (7.82)

34. Primary Outcome: Change in DL[CO] (% Predicted) From Baseline to EOS
Description: Change in DL[CO] (% predicted) from baseline to EOS were predicted. Extension baseline for safety is the last valid non-missing assessment that is taken on or after EOT visit in the core study, and prior to first study drug intake in the extension study.
Time Frame: as for outcome 31
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Percentage predicted DL[CO]
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 39 | 35
Percentage predicted DL[CO] | 9.3 (39.38) | 2.2 (49.50)

35. Other Pre Specified Outcome: Actual Values of 12-lead ECG Measurements on Day of First Re-initiation (Day 1) of Study Drug: Heart Rate
Description: Actual values of 12-lead ECG measurements on day of first Re-initiation (Day 1) of study drug: heart rate were reported.
Time Frame: Extension analysis period: Predose, 1, 2, 3, 4 hours post dose on Day 1 of re-initiation (re-initiation could occur on any day during the treatment period when drug was interrupted for at least 3 consecutive days [up to 71.8 months])
Population: Population analysis included numbers of participants based on sub-set of extension set who had a re-initiation. Here, 'n' (number analyzed) is defined as participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 30 | 40
beats per minute (bpm)
  Predose | 68.1 (8.73) | 71.0 (9.21)
  1 hour Post-dose: number analyzed (Participants) | 24 | 34
  1 hour Post-dose | 66.5 (10.53) | 69.0 (10.13)
  2 hours Post-dose: number analyzed (Participants) | 24 | 31
  2 hours Post-dose | 64.3 (9.91) | 65.1 (8.68)
  3 hours Post-dose: number analyzed (Participants) | 24 | 31
  3 hours Post-dose | 64.6 (9.33) | 67.8 (10.71)
  4 hours Post-dose: number analyzed (Participants) | 24 | 31
  4 hours Post-dose | 66.0 (9.73) | 67.6 (10.01)

36. Other Pre Specified Outcome: Actual Values of 12-lead ECG Measurements on Day of First Re-initiation (Day 1) of Study Drug: PR, QRS, QT, QTcB, QTcF
Description: Actual values of 12-lead ECG measurements on day of first Re-initiation (Day 1) of study drug: PR, QRS, QT, QTcB, QTcF were reported.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: millisecond (ms)
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
Number analyzed (Participants) | 30 | 40
millisecond (ms)
  PR Interval: Predose | 152.8 (17.66) | 149.8 (19.13)
  PR Interval: 1 hour Post-dose: number analyzed (Participants) | 24 | 34
  PR Interval: 1 hour Post-dose | 150.5 (17.25) | 152.6 (22.66)
  PR Interval: 2 hours Post-dose: number analyzed (Participants) | 24 | 31
  PR Interval: 2 hours Post-dose | 150.1 (16.60) | 153.6 (23.51)
  PR Interval: 3 hours Post-dose: number analyzed (Participants) | 24 | 31
  PR Interval: 3 hours Post-dose | 152.3 (17.73) | 154.5 (21.91)
  PR Interval: 4 hours Post-dose: number analyzed (Participants) | 24 | 31
  PR Interval: 4 hours Post-dose | 150.7 (17.82) | 151.8 (19.68)
  QRS Duration: Predose | 94.6 (11.06) | 91.5 (7.03)
  QRS Duration: 1 hour Post-dose: number analyzed (Participants) | 24 | 34
  QRS Duration: 1 hour Post-dose | 95.2 (11.42) | 93.2 (8.72)
  QRS Duration: 2 hours Post-dose: number analyzed (Participants) | 24 | 31
  QRS Duration: 2 hours Post-dose | 93.9 (11.71) | 92.7 (7.57)
  QRS Duration: 3 hours Post-dose: number analyzed (Participants) | 24 | 31
  QRS Duration: 3 hours Post-dose | 94.5 (11.60) | 94.5 (7.80)
  QRS Duration: 4 hours Post-dose: number analyzed (Participants) | 24 | 31
  QRS Duration: 4 hours Post-dose | 94.7 (10.48) | 92.5 (7.35)
  QT Interval: Predose | 391.5 (24.80) | 378.8 (23.61)
  QT Interval: 1 hour Post-dose: number analyzed (Participants) | 24 | 34
  QT Interval: 1 hour Post-dose | 396.7 (28.76) | 380.9 (21.78)
  QT Interval: 2 hours Post-dose: number analyzed (Participants) | 24 | 31
  QT Interval: 2 hours Post-dose | 402.0 (29.00) | 386.0 (19.62)
  QT Interval: 3 hours Post-dose: number analyzed (Participants) | 24 | 31
  QT Interval: 3 hours Post-dose | 400.2 (27.78) | 386.9 (21.38)
  QT Interval: 4 hours Post-dose: number analyzed (Participants) | 24 | 31
  QT Interval: 4 hours Post-dose | 400.0 (27.49) | 383.9 (23.14)
  QTcB Interval: Predose | 416.2 (19.05) | 411.4 (20.85)
  QTcB Interval: 1 hour Post-dose: number analyzed (Participants) | 24 | 34
  QTcB Interval: 1 hour Post-dose | 416.0 (24.11) | 407.6 (22.96)
  QTcB Interval: 2 hours Post-dose: number analyzed (Participants) | 24 | 31
  QTcB Interval: 2 hours Post-dose | 414.8 (22.83) | 401.7 (20.88)
  QTcB Interval: 3 hours Post-dose: number analyzed (Participants) | 24 | 31
  QTcB Interval: 3 hours Post-dose | 414.2 (23.30) | 410.1 (22.33)
  QTcB Interval: 4 hours Post-dose: number analyzed (Participants) | 24 | 31
  QTcB Interval: 4 hours Post-dose | 418.0 (20.30) | 406.6 (22.33)
  QTcF Interval: Predose | 407.4 (17.09) | 400.0 (18.69)
  QTcF Interval: 1 hour Post-dose: number analyzed (Participants) | 24 | 34
  QTcF Interval: 1 hour Post-dose | 409.2 (20.58) | 398.1 (18.22)
  QTcF Interval: 2 hours Post-dose: number analyzed (Participants) | 24 | 31
  QTcF Interval: 2 hours Post-dose | 410.1 (20.41) | 396.2 (16.61)
  QTcF Interval: 3 hours Post-dose: number analyzed (Participants) | 24 | 31
  QTcF Interval: 3 hours Post-dose | 409.0 (20.97) | 402.0 (16.82)
  QTcF Interval: 4 hours Post-dose: number analyzed (Participants) | 24 | 31
  QTcF Interval: 4 hours Post-dose | 411.5 (18.36) | 398.5 (18.27)

ADVERSE EVENTS:
Time Frame: Serious and Other AEs:From treatment start in extension study to EOT+15 days in extension study. Actual time varied till 71.8 months+15 days; All-cause mortality:From extension study baseline to EOS in extension study. Actual time varied till 73.2 months
Description: The extension set included all participants who signed an informed consent to enter the extension study and who received at least one dose of ponesimod study medication in the extension study.
Arm/Group | Ponesimod 20 mg (Core and Extension Study) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension)
All-Cause Mortality (participants affected / at risk) | 1/439 | 0/438
Serious Adverse Events (participants affected / at risk) | 56/439 | 57/438
Other Adverse Events (participants affected / at risk) | 339/439 | 328/438
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ponesimod 20 mg (Core and Extension Study) (N=439) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension) (N=438)
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 1 | 0
Sinus Node Dysfunction (Cardiac disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Vertigo Positional (Ear and labyrinth disorders) | 1 | 0
Macular Oedema (Eye disorders) | 0 | 1
Vision Blurred (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Anal Fissure (Gastrointestinal disorders) | 1 | 0
Chronic Gastritis (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Functional Gastrointestinal Disorder (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Umbilical Hernia (Gastrointestinal disorders) | 0 | 2
Papillitis (General disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Hepatic Cytolysis (Hepatobiliary disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 3 | 3
Bronchitis (Infections and infestations) | 1 | 0
Complicated Appendicitis (Infections and infestations) | 2 | 0
Covid-19 (Infections and infestations) | 2 | 1
Covid-19 Pneumonia (Infections and infestations) | 1 (1) | 2
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 0
Hepatitis E (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 1
Large Intestine Infection (Infections and infestations) | 0 | 1
Meningitis Viral (Infections and infestations) | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Pyelonephritis Acute (Infections and infestations) | 0 | 1
Pyelonephritis Chronic (Infections and infestations) | 0 | 1
Respiratory Syncytial Virus Infection (Infections and infestations) | 1 | 0
Staphylococcal Abscess (Infections and infestations) | 1 | 0
Suspected Covid-19 (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Incarcerated Incisional Hernia (Injury, poisoning and procedural complications) | 1 | 0
Ligament Injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0
Meniscus Injury (Injury, poisoning and procedural complications) | 0 | 1
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 0 | 1
Tendon Injury (Injury, poisoning and procedural complications) | 1 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 2
Wrist Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Ankylosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Instability (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Amnesia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysaesthesia (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Hemianopia (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Migraine with Aura (Nervous system disorders) | 1 | 0
Multiple Sclerosis Relapse (Nervous system disorders) | 1 | 2
Partial Seizures with Secondary Generalisation (Nervous system disorders) | 0 | 1
Sacral Radiculopathy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 1 | 1
Uhthoff's Phenomenon (Nervous system disorders) | 0 | 1
Vertigo CNS Origin (Nervous system disorders) | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Unintended Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Device Dislocation (Product Issues) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Mental Disorder Due to A General Medical Condition (Psychiatric disorders) | 0 | 1
Mood Disorder Due to A General Medical Condition (Psychiatric disorders) | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 0 | 1
Calculus Urinary (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal Colic (Renal and urinary disorders) | 2 | 0
Tubulointerstitial Nephritis (Renal and urinary disorders) | 2 | 1
Cervical Dysplasia (Reproductive system and breast disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 1 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0
Uterine Polyp (Reproductive system and breast disorders) | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominoplasty (Surgical and medical procedures) | 0 | 1
Abortion Induced (Surgical and medical procedures) | 2 | 1
Botulinum Toxin Injection (Surgical and medical procedures) | 0 | 1
Cervical Conisation (Surgical and medical procedures) | 0 | 1
Hysterosalpingo-Oophorectomy (Surgical and medical procedures) | 0 | 1
Inguinal Hernia Repair (Surgical and medical procedures) | 1 | 0
Internal Fixation of Fracture (Surgical and medical procedures) | 0 | 1
Mastectomy (Surgical and medical procedures) | 1 | 0
Osteotomy (Surgical and medical procedures) | 0 | 1
Spinal Operation (Surgical and medical procedures) | 1 | 0
Uterine Dilation and Curettage (Surgical and medical procedures) | 1 | 1
Uvulopalatopharyngoplasty (Surgical and medical procedures) | 0 | 1
Iliac Artery Embolism (Vascular disorders) | 1 | 0
Peripheral Artery Thrombosis (Vascular disorders) | 1 | 0
Varicose Vein (Vascular disorders) | 1 | 0
Venous Thrombosis Limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ponesimod 20 mg (Core and Extension Study) (N=439) | Teriflunomide 14 mg (Core) Then Ponesimod 20 mg (Extension) (N=438)
Leukopenia (Blood and lymphatic system disorders) | 18 | 23
Lymphopenia (Blood and lymphatic system disorders) | 66 | 64
Diarrhoea (Gastrointestinal disorders) | 22 | 15
Fatigue (General disorders) | 24 | 30
Covid-19 (Infections and infestations) | 115 | 108
Nasopharyngitis (Infections and infestations) | 82 | 74
Respiratory Tract Infection (Infections and infestations) | 23 | 15
Upper Respiratory Tract Infection (Infections and infestations) | 47 | 51
Urinary Tract Infection (Infections and infestations) | 36 | 33
Alanine Aminotransferase Increased (Investigations) | 73 | 98
Aspartate Aminotransferase Increased (Investigations) | 17 | 26
Lymphocyte Count Decreased (Investigations) | 30 | 30
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 | 38
Back Pain (Musculoskeletal and connective tissue disorders) | 45 | 30
Dizziness (Nervous system disorders) | 22 | 17
Headache (Nervous system disorders) | 57 | 64
Hypertension (Vascular disorders) | 37 | 44

LIMITATIONS AND CAVEATS:
Due to limited availability of COVID-19 vaccine-naïve MS patients, the COVID-19 vaccination sub-study was cancelled and removed from the protocol after implementation of amendment 5.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT03232073/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-04): https://cdn.clinicaltrials.gov/large-docs/73/NCT03232073/SAP_001.pdf